CLINICAL TRIAL: NCT06811935
Title: Feasibility of a Study to Determine the Incidence and Natural History of Children With Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS)
Brief Title: PEDI Pediatric Autoimmune Neuropsychiatric Disorder Associated With Streptococcus Study
Acronym: PANDAS
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2024-1009; Protocol Version 11/6/2025 (Other: UW Madison); A536756 (Other: UW Madison); 1R21MH138881-01 (NIH)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: PANS; PANDAS
MeSH Terms: conditions — Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — When possible, a research only blood sample will be collected, and serum will be saved for future use and possible sharing (In Primary Care participants only). This blood sample will be spun down and the serum separated and stored in a freezer. There will not be genetic testing done on this or any sample collected in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with PANS or PANDAS: This cohort will include participants from an In Primary Care Group where the patient is a current member of the primary care population at either UW Health or Dartmouth Health and an External to Primary Care Group.

SUMMARY:
The objective of the Pediatric Epidemiological Data and Incidence (PEDI) PANDAS study is to demonstrate the feasibility of enrollment and retention of subjects in a study to determine the incidence and natural history of children with Pediatric Acute-Onset Neuropsychiatric Syndrome (PANS) with regard to spectrum, course and outcome. The investigators aim to demonstrate they can recruit and retain 85% of children who are eligible for this study. Eligible children are those who fit criteria for PANS and Pediatric Autoimmune Neuropsychiatric Disorder Associated with Streptococcus (PANDAS). Each child will be followed for one year.

DETAILED DESCRIPTION:
Specific Aim 1: To establish proof-of-concept of prospectively determining the incidence of PANDAS/PANS and the role of Group A streptococcus (GAS) in this group of disorders.

Specific Aim 1a: To prospectively identify and enroll children with PANDAS and PANS in geographically distinct populations of children in the US in order to determine the incidence and spectrum of these disorders.

Specific Aim 1b: To determine the role of GAS in new onset PANDAS/PANS.

Specific Aim 2a: To establish proof-of-concept for studying the clinical course and outcome over the first year of treatment prospectively in children identified through the EHR in a primary care population.

Specific Aim 2b: To augment the number of children identified and establish proof-of-concept for studying the clinical course and outcome over the first year of treatment. Investigators will prospectively enroll children recently diagnosed with PANDAS/PANS in our local specialty clinics (not included within our primary care population) within four months of symptom onset.

ELIGIBILITY:
Inclusion Criteria (All participants):

* Child age 3-17 years old
* Child and their parent/guardian are able to complete all study activities in English
* Potential participant's family plans to be followed within UW Health or Dartmouth Health for at least one year

Inclusion Criteria (In primary care group only):

* Pediatric patient who is a current member of the primary care population at either UW Health or Dartmouth Health
* Abrupt onset of symptoms (within 7 days) occurring in the past 3 months. Willing to come in-person for at least the baseline visit.
* Suspected diagnosis of PANS or PANDAS based on published criteria:

  * PANS: (A) Abrupt, dramatic, overnight onset of obsessive compulsive disorder (OCD) or severely restricted food intake; (B) concurrent abrupt onset of additional severe neuropsychiatric symptoms from at least 2 of the following 7 categories:

    1. Anxiety
    2. Emotional lability and/or depression
    3. Irritability, aggression and/or severe oppositional behaviors
    4. Developmental regression
    5. Deterioration in school performance
    6. Sensory or motor abnormalities, including heightened sensitivity to sensory stimuli, hallucinations, dysgraphia, complex motor, and/or vocal tics
    7. Somatic signs and symptoms, including sleep disturbances, enuresis or urinary frequency consistent with a known neurologic or medical disorder.

AND (C) symptoms not better explained by another medical or neurologic disorder

* PANDAS

  * Presence of OCD and/or tic disorder
  * Pre-pubertal onset of symptoms (i.e., 3-12 years old)
  * Episodic course characterized by very acute and severe onset and dramatic symptom exacerbations
  * Neurologic abnormalities present during symptom exacerbations-motoric hyperactivity and adventitious movements
  * Temporal relationships between group A streptococcus (GAS) infections and symptom exacerbations

Inclusion Criteria - External to Primary Care Group ONLY:

* Abrupt onset of symptoms (within 7 days) occurring in the past 4 months.
* Confirmed diagnosis of PANS or PANDAS based on published criteria (see above).

Exclusion Criteria (all participants):

* History of tics, OCD or food restriction/avoidance that contradicts a history of sudden onset or was present before the onset of this investigation
* Current symptom(s) of Pica
* Previous participation in the study
* Not suitable for study participation at the discretion of the site investigator (e.g., the child does not have verbal or cognitive ability adequate for self-report assessment)
* Patient or family is unable to complete the study questionnaires or procedures in English as the primary language

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between the ages of 3 and 17 years with PANS or PANDAS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Eligible Participants Enrolled | up to 12 months
  To demonstrate that the methods of recruitment are effective, the aim is to enroll 85 percent of children with PANS/PANDAS who meet preliminary eligibility criteria for the study.

SECONDARY OUTCOMES:
Percentage of Participants Retained at 12 months | up to 12 months
  The secondary endpoint is retention in the study. The investigators hypothesize that at the 12-month visit, 85 percent of the children who are enrolled will still be on study.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Wald, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (2):
- United States (2):
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - UW School of Medicine and Public Health, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes